CLINICAL TRIAL: NCT00371826
Title: A Prospective, Open-label, Controlled Multicenter Trial to Assess the Efficacy and Safety of an Induction Regimen of Cyclosporine Micro Emulsion, Enteric-coated Mycophenolate Sodium (EC-MPS) and Corticosteroids, Followed by Administration of Everolimus and Enteric-coated Mycophenolate Sodium (EC-MPS), With Either the Withdrawal of Cyclosporine Micro Emulsion or Corticosteroids in de Novo Kidney Transplant Recipients
Brief Title: SOCRATES: Steroid or Cyclosporine Removal After Transplantation Using Everolimus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001A2421
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-06

CONDITIONS: Renal Transplanted Recipients
Keywords: Renal transplantation; everolimus; Immunosuppressants
MeSH Terms: interventions — Everolimus; Cyclosporine; Calcineurin Inhibitors; cni protein, Drosophila; Prednisone; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Calcineurin Inhibitor (CNI) Withdrawal (Experimental): Every randomized patient in this group received
  Day 1 - Day 14: cyclosporine as Calcineurin Inhibitor (CNI) 5 mg/kg twice daily (b.i.d.), dose adjusted to achieve C2 target of 1,500 ng/mL (range 1,400-1,600 ng/mL) + mycophenolate sodium (MPA)720 mg b.i.d. + methylprednisone/prednisone 500 mg intra-operatively, 250 mg on day 1, then 10-30 mg/day prednisone
  Day 15 - Day 60: everolimus 1.5 mg b.i.d. to achieve target 6-10 ng/mL + cyclosporine decrease dose as per protocol guideline + MPA 720 mg b.i.d. until everolimus trough >6 ng/mL, then MPA was stopped + prednisone 10-30mg/day
  Day 61 - Day 120: everolimus dose adjusted to achieve target 6-10 ng/mL + cyclosporine 25% dose reduction per fortnight, to be discontinued by day 120 as per protocol (or commence reduction by day 120 at discretion of investigator, to be completed within 2 months of commencement) + prednisone 10-30mg/day Day 121 - Month 36: everolimus dose adjusted to achieve target 8-12 ng/mL + prednisone 5-10 mg/day
  Interventions: Drug: Everolimus (RAD001); Drug: Cyclosporine (Calcineurin Inhibitor (CNI)); Drug: Methylprednisone/prednisone; Drug: Mycophenolate sodium (MPA)
- Steroid Withdrawal (Experimental): Every randomized patient in this group received
  Day 1 -14: cyclosporine 5 mg/kg b.i.d., dose adjusted to achieve C2 target as per protocol + mycophenolate sodium (MPA) 720 mg b.i.d. + methylprednisone/prednisone 500 mg intra-operatively, 250 mg on day 1, then 10-30 mg prednisone per day
  Day 15 - 60: everolimus 1.5 mg b.i.d. to achieve target 6-10 ng/mL + cyclosporine decrease dose as per protocol guideline + MPA 720 mg b.i.d. until everolimus trough >6 ng/mL, then MPA was stopped + prednisone 10-30mg per day
  Day 61 - 120: Everolimus dose adjusted + cyclosporine adjust dose according protocol guideline (or commence reduction by day 120 at discretion of Investigator, to be completed within 2 months of commencement) + gradual withdrawal of prednisone by 1 mg/week to be discontinued by Day 120.
  Day 121 - Month 36: At Day 121, Month 7 and Month 13 Everolimus dose was adjusted to achieve target 6-10 ng/mL + Cyclosporine adjust dose to achieve C2 target as per protocol
  Interventions: Drug: Everolimus (RAD001); Drug: Cyclosporine (Calcineurin Inhibitor (CNI)); Drug: Methylprednisone/prednisone; Drug: Mycophenolate sodium (MPA)
- CNI+MPA+ Steroid (Active Comparator): Patients randomized to this group received:
  Day 1 - Month 36: cyclosporine 5 mg/kg b.i.d., dose adjusted to achieve the protocol defined C2 Targets + mycophenolate sodium 720mg b.i.d. + Methylprednisone/prednisone 500mg intra-operatively, 250mg on day 1, 10-30mg prednisone per day until month 12 (as per local practice), 5-10mg/day months 13-36.
  Interventions: Drug: Cyclosporine (Calcineurin Inhibitor (CNI)); Drug: Methylprednisone/prednisone; Drug: Mycophenolate sodium (MPA)

INTERVENTIONS:
Drug: Everolimus (RAD001)
  Other Names: Certican®
  Arms: Calcineurin Inhibitor (CNI) Withdrawal; Steroid Withdrawal
Drug: Cyclosporine (Calcineurin Inhibitor (CNI))
  Other Names: Neoral®
Drug: Methylprednisone/prednisone
Drug: Mycophenolate sodium (MPA)
  Other Names: myfortic®

SUMMARY:
The aim of this study is to assess the safety and efficacy of corticosteroid discontinuation versus cyclosporine micro emulsion discontinuation in recipients receiving reduced exposure cyclosporine micro emulsion and corticosteroids plus enteric-coated mycophenolate sodium (EC-MPS) initially, changed to everolimus at 2 weeks post-transplant. These two groups will be compared to a third control group, who will receive treatment consisting of cyclosporine micro emulsion, enteric-coated mycophenolate sodium (EC-MPS) and steroids.

ELIGIBILITY:
Inclusion criteria

1. Males and females aged 18-65 years inclusive.
2. First time recipients of cadaveric, living unrelated or living related donor kidney transplants.
3. Patients who are willing and able to participate in the study and from whom written informed consent has been obtained.

Exclusion criteria

1. Patients who are recipients of multiple organ transplants, including more than one kidney, kidney and pancreas, or previous transplant with any organ other than kidney.
2. Patients at high immunological risk of graft loss, indicated by peak PRA >50% or loss of a previous renal allograft within the first 6 months of transplantation due to acute rejection.
3. Patients who have received an investigational drug within 4 weeks prior to the screening visit.
4. Presence of any severe allergy or hypersensitivity to drugs similar to everolimus (e.g. antibiotics such as Clindamycin)

Other protocol-defined inclusion/exclusion criteria may applied

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2006-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (7):
- Australia (7):
  - Royal Prince Alfred Hospital, NSW
  - Westmead Hospital, NSW
  - Princess Alexandra Hospital, QLD
  - Monash Medical Centre, Sale
  - Queen Elizabeth Hospital, Sale
  - Royal Melbourne Hospital, VIC
  - Sir Charles Gairdner Hospital, WA

RESULTS

PARTICIPANT FLOW:
Period: Core Phase (12 Months)
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Started | 49 ("Started" indicates patients in Randomized, Intent to treat (ITT) and Safety set.) | 47 | 30
Modified Intent to Treat (mITT)- Add | 46 | 44 | 20
Modified Intent to Treat (mITT) | 27 | 39 | 6
Completed | 25 ("Completed" means patients were still on study medication by month 12.) | 39 | 6
Not Completed | 24 | 8 | 24
Not completed — Adverse Event | 15 | 4 | 9
Not completed — Abnormal test procedure result(s) | 1 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 6 | 3 | 2
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Subject withdrew consent | 0 | 0 | 3
Not completed — Administrative problems | 1 | 0 | 8
Not completed — Graft Loss | 0 | 1 | 0
Period: Extension Phase (24 Months)
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Started | 23 (2 patients who completed 12 month core did not wish to continue in extension.) | 39 | 5 (One patient completed core, did not wish to continue to extension.)
Intention to Treat - Extenstion (ITT-Ex) | 23 | 39 | 4 (One patient entered extension, was withdrawn (no efficacy data in extension) due to DMC suggestion)
Safety Set | 22 (One patient randomized to this arm, was treated with the control regimen (CNI+MPA+Steroid)) | 40 (One patient mis-randomised to 1st arm but treated in this arm, evaluated for safety in this arm.) | 5 (Patient withdrawn as per DMC suggestion had no efficacy data, but was included in safety set.)
Completed | 18 | 29 | 3
Not Completed | 5 | 10 | 2
Not completed — Adverse Event | 4 | 5 | 0
Not completed — Abnormal test procedure result(s) | 0 | 1 | 0
Not completed — Unsatisfactory therapeutic effect | 0 | 2 | 0
Not completed — Subject withdrew consent | 1 | 2 | 0
Not completed — Administrative problems | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal | Total
Number analyzed (Participants) | 49 | 47 | 30 | 126
Age Continuous [Mean (Standard Deviation); unit: years] | 48.4 (10.17) | 45.8 (10.83) | 43.5 (10.66) | 46.3 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 6 | 36
  Male | 32 | 34 | 24 | 90

OUTCOME MEASURES:

1. Primary Outcome: Calculated Glomerular Filtration Rate (cGFR) After Kidney Transplant to Evaluate Kidney Function (12 Months Analysis)
Description: The glomerular filtration rate (GFR) was calculated by the Nankivell formula: GFR = 6.7 / Scr + BW / 4 - Surea / 2-100 / (height)^ 2 + C where Scr is the serum creatinine concentration expressed in mmol/L, BW the body weight in kg, Surea the serum urea in mmol/L, height in m, and the constant C is 35 for male and 25 for female patients.
Time Frame: At Month 12
Population: Modified intent-to-treat (mITT)-Add population: All ITT patients who had a calculated GFR value recorded at Month 12 post-randomization including those collected after discontinuation of study medication and retrospectively collected creatinine and urea data
Measure: Mean (Standard Deviation); unit: mL/min per 1.73 m^2
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 46 | 44 | 20
mL/min per 1.73 m^2 | 65.2 (15.52) | 69.3 (15.18) | 66.9 (16.22)

2. Secondary Outcome: Calculated Glomerular Filtration Rate (cGFR) After Kidney Transplant to Evaluate Kidney Function (36 Months Analysis)
Description: as for outcome 1
Time Frame: At Month 24 and 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period. Missing values were imputed by last observation carried forward (LOCF) using values beyond Month 6
Measure: Mean (Standard Error); unit: mL/min per 1.73 m^2
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 36 | 4
mL/min per 1.73 m^2
  Month 24 (n= 23, 36, 4) | 69.5 (12.60) | 71.8 (16.37) | 67.0 (14.72)
  Month 36 (n= 19, 35, 3) | 71.6 (17.50) | 69.1 (14.77) | 61.0 (11.36)

3. Secondary Outcome: Number of Participants With Biopsy Proven Acute Rejection (BPAR) Per Treatment Group (12 Months Analysis)
Description: A biopsy-proven acute rejection is defined as a biopsy graded IA, IB, IIA, IIB, or III as per Banff 97 classification.
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population: All patients who were randomized. This population also included all patients who were randomized but were not treated with study medication.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants | 15 | 6 | 5

4. Secondary Outcome: Number of Participants With Biopsy Proven Acute Rejection (BPAR) Per Treatment Group (36 Months Analysis)
Description: A biopsy-proven acute rejection is defined as a biopsy graded IA, IB, IIA, IIB, or III as per Banff 97 classification.
Time Frame: At Month 12, 24 and 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period. This population includes also all patients who were randomized but were not treated with study medication.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  At Month 12 | 4 | 4 | 0
  At Month 24 | 5 | 5 | 0
  At Month 36 | 6 | 8 | 0

5. Secondary Outcome: Number of Participants With Composite Endpoint of Treatment Failure (12 Months Analysis)
Description: Composite endpoint of treatment failure includes biopsy-proven acute rejection (BPAR), graft loss, death and loss-to-follow-up. A BPAR is defined as a biopsy graded IA, IB, IIA, IIB, or III as per Banff 97 classification.
  The allograft was presumed to be lost on the day the patient started dialysis and was not able to subsequently be removed from dialysis. If the patient underwent a graft nephrectomy, then the day of nephrectomy was the day of graft loss.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants | 16 | 8 | 11

6. Secondary Outcome: Number of Participants With Composite Endpoint of Treatment Failure (36 Months Analysis)
Description: as for outcome 5
Time Frame: At Month 12, 24 and 36
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  At Month 12 | 4 | 4 | 0
  At Month 24 | 6 | 6 | 0
  At Month 36 | 7 | 10 | 0

7. Secondary Outcome: Number of Participants With Histological Evidence Chronic Allograft Nephropathy (CAN) (12 Months Analysis)
Description: A per-protocol biopsy was performed at Baseline and Month 12 and read by an independent blinded pathologist in order to assess chronic allograft nephropathy. Chronic rejection is characterized by a slow progressive decline in renal function and is typically preceded by the histological picture of chronic allograft nephropathy. The presence of biopsy confirmed Grade I, II or III chronic allograft nephropathy by Banff 97 criteria was assessed on all optional biopsies obtained for clinical suspicion of chronic rejection.
  Data summarized by 3 categories. "Yes" - Patients with histological evidence of CAN ; "No" - Patients with histological evidence of CAN and "Not Done" - Central protocol defined kidney allograft biopsies were not done.
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population: All patients who were randomized. This population also included all patients who were randomized but were not treated with study medication. For this analysis, only patients with available data were included. The analysis included biopsies of Month 12 visit that were done beyond month 12 cut-off date.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 30 | 40 | 10
Participants
  YES | 8 | 6 | 2
  NO | 15 | 26 | 5
  Not Done | 7 | 8 | 3

8. Secondary Outcome: Number of Participants With Histological Evidence Chronic Allograft Nephropathy (CAN) (36 Months Analysis)
Description: Chronic rejection is characterized by a slow progressive decline in renal function and is typically preceded by the histological picture of chronic allograft nephropathy. The presence of biopsy confirmed Grade I, II or III chronic allograft nephropathy by Banff 97 criteria was assessed on all optional biopsies obtained for clinical suspicion of chronic rejection.
  Data summarized by 3 categories. "Yes" - Patients with histological evidence of CAN ; "No" - Patients with histological evidence of CAN and "Not Done" - Central protocol defined kidney allograft biopsies were not done.
Time Frame: At Month 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period. Patients with data available at month 36 were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 18 | 31 | 3
Participants
  YES | 2 | 1 | 1
  NO | 8 | 16 | 1
  Not Done | 8 | 14 | 1

9. Secondary Outcome: Number of Participants With Sub Clinical Acute Rejection (12 Months Analysis)
Description: Based on Banff 97 criteria, sub clinical acute rejection can be:
  GRADE IA - Cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  GRADE IB - Cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>10 mononuclear cells/tubular cross section or group of 10 tubular cells).
  GRADE IIA - Cases with significant interstitial infiltration and mild to moderate intimal arteritis (v1).
  GRADE IIB - Cases with moderate to severe intimal arteritis comprising >25% of the luminal area (v2).
  GRADE III - Cases with "transmural" arteritis or fibrinoid change and necrosis of medial smooth muscle cells (v3).
  "Borderline" category is used when no intimal arteritis is present, but there are foci of mild tubulitis (1 to 4 mononuclear cells/tubular cross section).
Time Frame: At Month 12
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 30 | 40 | 10
Participants
  NO | 20 | 29 | 5
  Borderline | 2 | 2 | 2
  Grade IA | 1 | 0 | 0
  Grade IB | 0 | 1 | 0
  Grade IIA | 0 | 0 | 0
  Grade IIB | 0 | 0 | 0
  Grade III | 0 | 0 | 0
  Not Done | 7 | 8 | 3

10. Secondary Outcome: Number of Participants With Sub Clinical Acute Rejection (36 Months Analysis)
Description: Based on Banff 97 criteria, sub clinical acute rejection can be:
  GRADE IA - Cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>4 mononuclear cells/tubular cross section or group of 10 tubular cells).
  GRADE IB - Cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>10 mononuclear cells/tubular cross section or group of 10 tubular cells).
  GRADE IIA - Cases with significant interstitial infiltration and mild to moderate intimal arteritis (v1).
  GRADE IIB - Cases with moderate to severe intimal arteritis comprising >25% of the luminal area (v2).
  GRADE III - Cases with "transmural" arteritis or fibrinoid change and necrosis of medial smooth muscle cells (v3).
  "Borderline' category is used when no intimal arteritis is present, but there are foci of mild tubulitis (1 to 4 mononuclear cells/tubular cross section).
Time Frame: At Month 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 18 | 31 | 3
Participants
  Month 36: NO | 9 | 15 | 2
  Month 36: Borderline | 1 | 1 | 0
  Month 36: Grade IA | 0 | 1 | 0
  Month 36: Grade IB | 0 | 0 | 0
  Month 36: Grade IIA | 0 | 0 | 0
  Month 36: Grade IIB | 0 | 0 | 0
  Month 36: Grade III | 0 | 0 | 0
  Month 36: Not Done | 8 | 14 | 1

11. Secondary Outcome: Mean Serum Creatinine (12 Months Analysis)
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population: All patients who were randomized. This population also included all patients who were randomized but were not treated with study medication. Patients with 12 month data on serum creatinine were included in this analysis.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 33 | 43 | 11
umol/L | 118.9 (31.59) | 161.0 (169.22) | 148.6 (76.84)

12. Secondary Outcome: Mean Serum Creatinine (36 Months Analysis)
Time Frame: At Month 12, 18, 24 and 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period. Patients with data on creatinine serum creatinine were included in this analysis. Last observation carried forward (LOCF) imputation technique was used.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
umol/L
  At Month 12 (n= 23, 39, 4) | 112.7 (33.38) | 123.0 (33.10) | 146.8 (89.36)
  At Month 18 (n= 22, 36, 4) | 113.6 (34.56) | 121.4 (35.78) | 146.3 (89.16)
  At Month 24 (n = 23, 36, 4) | 119.9 (36.83) | 123.7 (35.20) | 146.5 (78.20)
  At Month 36 (n= 19, 35, 3) | 119.4 (47.50) | 131.8 (42.30) | 176.0 (87.28)

13. Secondary Outcome: Creatinine Clearance (CrCl) Calculated by the Cockcroft-Gault Formula (12 Months Analysis)
Description: Creatinine clearance were calculated according to the Cockcroft-Gault formula:
  CrCl (males) = (140-A) × BW/(72 × Cr) CrCl (females) = CrCl (males) × 0.85 where A is age [years], BW is body weight [kg], and Cr is the serum concentration of creatinine [mg/dL].
  The Cockcroft-Gault formula estimates creatinine clearance based on serum creatinine level, body weight, and age.
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population: All patients who were randomized. This population also included all patients who were randomized but were not treated with study medication. Patients with 12 month data on creatinine clearance were included in this analysis.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 33 | 43 | 11
mL/min | 66.1 (19.37) | 67.8 (21.85) | 63.2 (21.73)

14. Secondary Outcome: Creatinine Clearance Calculated by the Cockcroft-Gault Formula (36 Months Analysis)
Description: as for outcome 13
Time Frame: At Month 12, 24 and 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period. Patients with data on creatinine clearance were included in this analysis. Last observation carried forward (LOCF) imputation technique was used.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
mL/min
  At Month 12 (n= 23, 39, 4) | 69.8 (19.90) | 71.7 (17.68) | 63.7 (10.33)
  At Month 18 (n=22, 36, 4) | 69.9 (20.16) | 73.7 (19.34) | 66.2 (12.28)
  At Month 24 (n= 23, 36, 4) | 65.6 (18.83) | 72.8 (20.86) | 63.7 (5.76)
  At Month 36 (n= 23, 39, 4) | 66.3 (22.30) | 67.5 (16.01) | 62.7 (16.58)

15. Secondary Outcome: Mean Urine Albumin/Creatinine Ratio (ACR) as Measurement of Proteinuria (12 Months Analysis)
Description: Proteinuria is measured by spot morning urine Albumin/Creatinine Ratio [ACR]. When the ACR is more than or equal to 30 mg/mmol then it is known as proteinuria.
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population: All patients who were randomized. This population also included all patients who were randomized but were not treated with study medication. Patients with 12 month data on Proteinuria were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/mg
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 22 | 32 | 4
mg/mg | 0.2 (0.27) | 0.1 (0.12) | 0.1 (0.02)

16. Secondary Outcome: Mean Urine Albumin/Creatinine Ratio [ACR] as Measurement of Proteinuria (36 Months Analysis)
Description: as for outcome 15
Time Frame: At Month 12, 18, 24 and 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment in extension period. This also includes all patients who were randomized but were not treated with study medication. Patients with ACR data at particular time point were included for analysis.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 18 | 32 | 2
mg/mmol
  At 12 Month (n = 18, 32, 2) | 23.5 (31.51) | 8.1 (13.40) | 4.8 (3.80)
  At 18 Month (n= 17, 31, 2) | 28.2 (47.78) | 8.1 (12.00) | 5.3 (4.12)
  At 24 Month ( n= 16, 29, 1) | 30.0 (51.72) | 6.6 (14.69) | 7.0 (NA) — One patient data analyzed in this arm, hence no standard deviation available.
  At 36 Month ( n= 15, 25, 0) | 30.6 (40.18) | 23.4 (66.51) | NA (NA) — No patient, hence no data available.

17. Secondary Outcome: Number of Participants With Post Transplant Diabetes Mellitus (PTDM) and Impaired Fasting Glucose (12 Months Analysis)
Description: The symptoms of post transplant diabetes mellitus (PTDM) and impaired fasting glucose are defined as any of the following conditions:
  1. Patients receiving glucose lowering treatment
  2. Fasting plasma glucose (FPG) >= 126 mg/dL on 2 separate occasions
  3. Hemoglobin subtype A1c (HbA1c) > 6.5%
  4. Diabetes reported as treatment emergent AE with end date > Day 15
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population: All patients who were randomized. This population also included all patients who were randomized but were not treated with study medication. Patients with 12 month data on PTDM were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 38 | 42 | 25
Participants
  Glucose lowering treatment | 10 | 9 | 5
  FPG >= 126 mg/dL on 2 separate occasions | 6 | 0 | 5
  HbA1c > 6.5% | 12 | 3 | 5
  Diabetes as treatment emergent AE | 8 | 2 | 3
  Any of the above symptoms | 19 | 10 | 8

18. Secondary Outcome: Number of Participants With New Onset Diabetes Mellitus After Transplantation (NODAT) and Impaired Fasting Glucose (36 Months Analysis)
Description: The symptoms of new onset diabetes mellitus after transplantation (NODAT) and impaired fasting glucose are defined as any of the following conditions:
  1. Patients receiving glucose lowering treatment
  2. 2 fasting plasma glucose (FPG) values >= 126 mg/dL or 2 random plasma glucose (RPG) values >= 200 mg/dL or FPG value >= 126 mg/dL and 1 RPG value >= 200 mg/dL
  3. Diabetes reported as treatment emergent AE with end date > Day 15
Time Frame: At Month 36
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period. This also includes patients who were randomized but were not treated with study drug.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  Glucose lowering treatment | 5 | 10 | 2
  FPG or RPG | 3 | 2 | 1
  Diabetes as treatment emergent AE | 5 | 4 | 2
  Any of the above symptoms | 6 | 11 | 2

19. Secondary Outcome: Number of Participants With Notable Abnormal Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) as Measurement of Effect of Treatment on Cardiovascular Health (12 Months Analysis)
Description: Notable abnormal systolic blood pressure is defined as :
  * Either an increase of >=30 that results in >=180 or >200 (mm/Hg)
  * OR a decrease of >=30 that results in <=90 or <75 (mm/Hg)from baseline
  Notable abnormal diastolic blood pressure is defined as :
  * Either an increase of >=20 that results in >=105 or >115 (mm/Hg)
  * OR a decrease of >=20 that results in <=50 or <40 (mm/Hg) from baseline
Time Frame: Baseline, Overall post-baseline up to 12 month
Population: Safety population (SAF): All patients in whom transplantation was performed and who were treated with at least one dose of study medication and had at least one safety/tolerability assessment after randomization. Patients with baseline and overall post baseline up to 12 month assessment for this analysis were included.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants
  SBP: >=180 mm/Hg or 200 mm/Hg | 5 | 5 | 7
  SBP: < = 90 mm/Hg or < 200 mm/Hg | 1 | 0 | 0
  DBP : >=105 mm/Hg or >115 mm/Hg | 3 | 6 | 5
  DBP: <=50 mm/Hg or <40 mm/Hg | 1 | 4 | 0

20. Secondary Outcome: Number of Participants With Notable Abnormal Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) as Measurement of Effect of Treatment on Cardiovascular Health (36 Months Analysis)
Description: Notable abnormal systolic blood pressure is defined as :
  * Either an increase of >=30 that results in >=180 or >200 (mm/Hg)
  * OR a decrease of >=30 that results in <=90 or <75 (mm/Hg) from baseline
  Notable abnormal diastolic blood pressure is defined as :
  * Either an increase of >=20 that results in >=105 or >115 (mm/Hg)
  * OR a decrease of >=20 that results in <=50 or <40 (mm/Hg) from baseline
Time Frame: Baseline, Overall post baseline up to Month 36
Population: Safety population extension (SAF-EX): All patients who entered the extension period, treated with at least one dose of study medication during the extension period and had at least one safety/tolerability assessment after entering the extension period. Patients with baseline and overall post baseline up to month 36 assessment were included.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 22 | 40 | 5
Participants
  SBP: >=180 mm/Hg or 200 mm/Hg | 3 | 4 | 1
  SBP: < = 90 mm/Hg or < 200 mm/Hg | 1 | 0 | 0
  DBP : >=105 mm/Hg or >115 mm/Hg | 2 | 5 | 1
  DBP: <=50 mm/Hg or <40 mm/Hg | 1 | 4 | 0

21. Secondary Outcome: Number of Participants With Erythropoietin Usage (12 Months Analysis)
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
participants | 20 | 10 | 8

22. Secondary Outcome: Number of Participants With Erythropoietin Usage (36 Months Analysis)
Time Frame: Month 36
Population: as for outcome 18
Measure: Number; unit: participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
participants | 5 | 7 | 2

23. Secondary Outcome: Mean Short-form 36 Health Survey (SF-36) Score as a Measure of Quality of Life Assessment (12 Months Analysis)
Description: SF-36 measures impact of disease on overall quality of life (QoL). 36-item survey has 8 subscales. The 8 subscales are: Physical functioning (PF), Role-physical (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Role-emotional (RE) and Mental health (MH).
  Score for eash sub-scale has been standardized with the use of norm-based methods based on assessment of the general U.S. population free of chronic conditions. Scores range from 1-100 with a mean=50 and a standard deviation=10. A higher score indicates less impact on QoL.
Time Frame: At Month 12
Population: Intent-to-treat (ITT) population: All patients who were randomized. This population also included all patients who were randomized but were not treated with study medication. Only those patients who had completed the QoL assessment for Month 12 were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 24 | 37 | 5
units on a scale
  Physical functioning (PF) | 78.7 (26.53) | 76.9 (30.08) | 82.0 (34.93)
  Role-physical (RP) | 72.9 (40.99) | 78.2 (33.98) | 100.0 (0.00)
  Bodily pain (BP) | 73.6 (30.60) | 81.5 (19.21) | 96.8 (7.16)
  General health (GH) | 67.1 (22.41) | 71.2 (15.75) | 86.8 (12.91)
  Vitality (VT) | 62.7 (23.64) | 72.4 (15.88) | 85.0 (9.35)
  Social Functioning (SF) | 74.5 (30.72) | 81.1 (21.97) | 97.5 (5.59)
  Role-emotional (RE) | 72.2 (40.13) | 81.1 (34.73) | 100.0 (0.00)
  Mental health (MH) | 73.3 (21.02) | 79.1 (14.58) | 92.8 (7.69)

24. Secondary Outcome: Mean Short-form 36 Health Survey (SF-36) Score as a Measure of Quality of Life Assessment (36 Months Analysis)
Description: SF-36 measures impact of disease on overall quality of life (QoL). 36-item survey has 8 subscales. The 8 subscales are : Physical functioning (PF), Role-physical (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social functioning (SF), Role-emotional (RE) and Mental health (MH).
  Score for each sub-scale has been standardized with the use of norm-based methods based on assessment of the general U.S. population free of chronic conditions. Scores range from 1-100 with a mean=50 and a standard deviation=10. A higher score indicates less impact on QoL.
Time Frame: At Month 24
Population: Intent-to-treat population extension (ITT-EX): All patients who were randomized, entered the extension period, and had at least one efficacy assessment after entering the extension period. This also includes patients who were randomized but were not treated with study drug. Patients with completed SF-36 assessment were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 16 | 31 | 2
units on a scale
  Physical functioning (PF) | 84.3 (24.20) | 87.6 (17.70) | 90.0 (7.07)
  Role-physical (RP) | 75.0 (39.79) | 77.4 (33.76) | 100.0 (0.00)
  Bodily pain (BP) | 81.6 (20.57) | 85.0 (21.18) | 84.0 (0.00)
  General health (GH) | 71.6 (24.45) | 69.8 (16.46) | 67.0 (0.00)
  Vitality (VT) | 70.0 (23.59) | 72.7 (13.59) | 60.0 (14.14)
  Social Functioning (SF) | 85.9 (20.35) | 80.6 (23.46) | 68.8 (26.52)
  Role-emotional (RE) | 72.9 (30.35) | 83.9 (29.65) | 33.3 (0.00)
  Mental health (MH) | 77.5 (18.35) | 77.9 (16.37) | 62.0 (8.49)

25. Secondary Outcome: Number of Participants Hospitalized for Reasons Other Than Primary Transplantation (12 Months Analysis)
Description: This analysis is reporting number of participants hospitalized for reasons (such as acute rejection, infection, gastrointestinal (GI) events, cardiovascular event, metabolic disorder and Other) other than primary transplantation.
Time Frame: Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants | 34 | 31 | 13

26. Secondary Outcome: Number of Participants Hospitalized for Reasons Other Than Primary Transplantation (36 Months Analysis)
Description: as for outcome 25
Time Frame: Month 36
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants | 16 | 30 | 1

27. Secondary Outcome: Number of Participants With Employment Status (12 Months Analysis)
Description: The various employment status reported are:
  * Employed/self employed full time
  * Employed part time
  * Unemployed
  * Homemaker
  * Volunteer
  * Permanently disabled
  * Non-permanently disable
  * Retired
  * Other
Time Frame: At screening (at day 0 +/- 7 days ), At Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants
  Screening visit: Employed/self employed full time | 18 | 21 | 9
  Month 12: Employed/self employed full time | 6 | 14 | 2
  Screening visit: Employed part time | 9 | 7 | 4
  Month 12: Employed part time | 3 | 5 | 0
  Screening visit: Unemployed | 10 | 8 | 10
  Month 12: Unemployed | 6 | 1 | 6
  Screening visit: Homemaker | 3 | 5 | 5
  Month 12 : Homemaker | 2 | 5 | 2
  Screening visit: Volunteer | 1 | 0 | 0
  Month 12: Volunteer | 1 | 0 | 0
  Screening visit: Permanently disabled | 2 | 2 | 0
  Month 12: Permanently disabled | 1 | 2 | 0
  Screening visit: Non-permanently disabled | 1 | 2 | 0
  Month 12: Non-permanently disabled | 1 | 0 | 0
  Screening visit: Retired | 4 | 2 | 1
  Month 12: Retired | 1 | 2 | 0
  Screening visit: Other | 1 | 0 | 1
  Month 12: Other | 1 | 0 | 0

28. Secondary Outcome: Number of Participants With Employment Status (36 Months Analysis)
Description: as for outcome 27
Time Frame: At screening (at day 0 +/- 7 days ), At Month 36
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  Screening visit: Employed/self employed full time | 5 | 10 | 1
  Month 36: Employed/self employed full time | 4 | 10 | 1
  Screening visit: Employed part time | 4 | 7 | 0
  Month 36: Employed part time | 3 | 4 | 0
  Screening visit: Unemployed | 5 | 7 | 1
  Month 36: Unemployed | 3 | 6 | 0
  Screening visit: Homemaker | 3 | 3 | 1
  Month 36 : Homemaker | 3 | 3 | 1
  Screening visit: Permanently disabled | 0 | 1 | 0
  Month 36: Permanently disabled | 0 | 1 | 0
  Screening visit: Non-permanently disabled | 0 | 1 | 0
  Month 36: Non-permanently disabled | 0 | 1 | 0
  Screening visit: Retired | 0 | 2 | 0
  Month 36: Retired | 0 | 2 | 0
  Screening visit: Other | 1 | 0 | 0
  Month 36: Other | 1 | 0 | 0

29. Secondary Outcome: Number of Participants With Wound Problems(12 Months Analysis)
Description: Patients with any wound healing problem such as infection related to kidney surgery, dehiscence, lymphocele, hernia, seroma, hematoma, ureteral anastomotic complication and other were reported in this analysis.
Time Frame: At Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants
  Any wound healing problem | 16 | 15 | 9
  Infection related to kidney surgery | 2 | 4 | 3
  Dehiscence | 3 | 2 | 2
  Lymphocele | 3 | 4 | 3
  Hernia | 3 | 2 | 1
  Seroma | 4 | 9 | 3
  Hematoma | 4 | 0 | 2
  Ureteral anastomotic complication | 2 | 1 | 1
  Other | 3 | 1 | 0

30. Secondary Outcome: Number of Participants With Any Wound Problems (36 Months Analysis)
Description: as for outcome 29
Time Frame: At Month 12, 24 and 36
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  At Month 12 | 6 | 11 | 2
  At Month 24 | 9 | 13 | 2
  At Month 36 | 10 | 13 | 2

31. Secondary Outcome: Number of Participants With Notable Abnormalities in Total Cholesterol and Triglycerides as Measurement of Effect of Treatment on Cardiovascular Health (12 Months Analysis)
Description: Notable abnormal total cholesterol is defined as : High: >= 9.1 mmol/L , normal range is 0.00 - 5.17 mmol/L
  Notable abnormal triglycerides is defined as : High: >= 8.5 mmol/L, normal range is 0.30 - 2.00 mmol/L
Time Frame: Overall post baseline up to month 12
Population: Safety population (SAF): All patients in whom transplantation was performed and who were treated with at least one dose of study medication and had at least one safety/tolerability assessment after randomization. Patients with serum lipid assessment anytime post baseline up to 12 month were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 48 | 47 | 30
Participants
  Total Cholesterol: High (n = 48, 47,30) | 6 | 0 | 3
  Triglycerides : High (n= 48, 46, 30) | 1 | 0 | 0

32. Secondary Outcome: Number of Participants With Notable Abnormalities in Total Cholesterol and Triglycerides as Measurement of Effect of Treatment on Cardiovascular Health (36 Months Analysis)
Description: as for outcome 31
Time Frame: Overall Post Baseline up to month 36
Population: Safety population extension (SAF-EX): All patients who entered the extension period, treated with at least one dose of study medication during the extension period and had at least one safety/tolerability assessment after entering the extension period. Patients with serum lipid assessment anytime post baseline up to 36 month were included .
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 22 | 40 | 5
Participants
  Total Cholesterol: High | 6 | 0 | 1
  Triglycerides : High | 0 | 1 | 0

33. Secondary Outcome: Number of Participants With Antibody-mediated Rejection Per Treatment Group (12 Months Analysis)
Time Frame: At Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants | 5 | 2 | 2

34. Secondary Outcome: Number of Participants With Antibody-mediated Rejection Per Treatment Group (36 Months Analysis)
Time Frame: At Month 12, 24 and 36
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  At Month 12 | 1 | 0 | 0
  At Month 24 | 1 | 0 | 0
  At Month 36 | 1 | 2 | 0

35. Secondary Outcome: Number of Participants With Biopsy Proven Acute Rejection (BPAR) Influenced by Demographic Characteristics and Morbidities (12 Months Analysis)
Description: The influence of demographic characteristics and comorbidities on incidence of BPAR were analyzed in the following way: Demographic characteristics were age (<55 years, ≥55 years), Expanded criteria Donor (ECD) organ (donor age >60 years or donor non heart-beating and donor age >50), gender, living vs. deceased donor, Body Mass Index (BMI) classes (underweight <18.5, normal 18.5 - <25.0, overweight 25.0 - <30.0, obesity 30.0 and above), years on dialysis before transplantation (<1, 1-5, >5 years). Comorbidities were diabetes, hypertension, cardiovascular diseases/events, nephrosclerosis, glomerulonephritis/glomerular disease, polycystic disease, and Cytomegalovirus status.
Time Frame: At Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants
  Age < 55 years | 11 | 5 | 4
  Age > = 55 years | 4 | 1 | 1
  ECD Organ | 3 | 0 | 2
  NO ECD Organ | 12 | 6 | 3
  Male | 11 | 6 | 4
  Female | 4 | 0 | 1
  Living donor | 9 | 6 | 2
  Deceased donor | 6 | 0 | 3
  BMI < 18.5 | 0 | 1 | 0
  BMI 18.5 - <25 | 5 | 2 | 3
  BMI 25 - <30 | 8 | 3 | 1
  BMI >= 30 | 2 | 0 | 1
  Years on dialysis before transplantation: None | 1 | 0 | 0
  < 1 Year on dialysis before transplantation | 3 | 3 | 1
  1 - 5 Years on dialysis before transplantation | 8 | 1 | 2
  > 5 Years on dialysis before transplantation | 3 | 2 | 2
  Diabetes mellitus: No | 10 | 4 | 4
  Diabetes mellitus: Yes | 5 | 2 | 1
  Hypertension: No | 2 | 1 | 0
  Hypertension: Yes | 13 | 5 | 5
  Cardiovascular disease : No | 4 | 3 | 2
  Cardiovascular disease: Yes | 11 | 3 | 3
  Nephrosclerosis: No | 15 | 6 | 4
  Nephrosclerosis: Yes | 0 | 0 | 1
  Glomerulonephritis/glomerular disease : No | 8 | 5 | 3
  Glomerulonephritis/glomerular disease: Yes | 7 | 1 | 2
  Cytomegalovirus : Negative | 2 | 2 | 0
  Cytomegalovirus : Positive | 13 | 4 | 5

36. Secondary Outcome: Number of Participants With Biopsy Proven Acute Rejection (BPAR) Influenced by Demographic Characteristics and Morbidities (36 Months Analysis)
Description: The influence of demographic characteristics and comorbidities on incidence of BPAR were analyzed in the following way: Demographic characteristics were age (<55 years, ≥55 years), Expanded Criteria Donor [ECD] organ (donor age >60 years or donor non heart-beating and donor age >50), gender, living vs. deceased donor, Body Mass Index (BMI) classes (underweight <18.5, normal 18.5 - <25.0, overweight 25.0 - <30.0, obesity 30.0 and above), years on dialysis before transplantation (<1, 1-5, >5 years). Comorbidities were diabetes, hypertension, cardiovascular diseases/events, nephrosclerosis, glomerulonephritis/glomerular disease, polycystic disease, and Cytomegalovirus status.
Time Frame: At Month 36
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  Age < 55 years | 6 | 7 | 0
  Age > = 55 years | 0 | 1 | 0
  ECD Organ | 0 | 0 | 0
  NO ECD Organ | 6 | 8 | 0
  Male | 4 | 7 | 0
  Female | 2 | 1 | 0
  Living donor | 5 | 6 | 0
  Deceased donor | 1 | 2 | 0
  BMI < 18.5 | 1 | 0 | 0
  BMI 18.5 - <25 | 1 | 3 | 0
  BMI 25 - <30 | 4 | 4 | 0
  BMI >= 30 | 0 | 1 | 0
  Years on dialysis before transplantation: None | 0 | 1 | 0
  < 1 Year on dialysis before transplantation | 3 | 4 | 0
  1 - 5 Years on dialysis before transplantation | 2 | 2 | 0
  > 5 Years on dialysis before transplantation | 1 | 1 | 0
  Diabetes mellitus: No | 3 | 6 | 0
  Diabetes mellitus: Yes | 3 | 2 | 0
  Hypertension: No | 1 | 1 | 0
  Hypertension: Yes | 5 | 7 | 0
  Cardiovascular disease : No | 3 | 5 | 0
  Cardiovascular disease: Yes | 3 | 3 | 0
  Nephrosclerosis: No | 6 | 7 | 0
  Nephrosclerosis: Yes | 0 | 1 | 0
  Glomerulonephritis/glomerular disease : No | 4 | 7 | 0
  Glomerulonephritis/glomerular disease: Yes | 2 | 1 | 0
  Cytomegalovirus : Negative | 1 | 4 | 0
  Cytomegalovirus : Positive | 5 | 4 | 0

37. Secondary Outcome: Number of Patient Survival and Graft Survival (12 Months Analysis)
Time Frame: At Month 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 49 | 47 | 30
Participants
  Patient Survival | 49 | 46 | 30
  Graft Survival | 49 | 45 | 30

38. Secondary Outcome: Number of Patient Survival and Graft Survival (36 Months Analysis)
Time Frame: At Month 12, 24 and 36
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 23 | 39 | 4
Participants
  Month 12: Patient Survival | 23 | 39 | 4
  Month 12: Graft Survival | 23 | 39 | 4
  Month 24: Patient Survival | 23 | 39 | 4
  Month 24: Graft Survival | 23 | 39 | 4
  Month 36: Patient Survival | 23 | 39 | 4
  Month 36: Graft Survival | 23 | 39 | 4

39. Secondary Outcome: Change in Bone Mineral Density Between Week 2 and Month 24 (36 Months Analysis)
Description: Measurements of bone mineral density (BMD) by Dual Energy X-ray Absorptiometry (DEXA) were done at Week 2 and Month 24. Change in BMD between week 2 and Month 24 were done for neck of femur and lumbar spine.
Time Frame: Week 2, Month 24
Population: Safety population extension (SAF-EX): All patients who entered the extension period, who were treated with at least one dose of study medication during the extension period and had at least one safety/tolerability assessment after entering the extension period. Patients with week 2 and month 24 assessment for this analysis were included.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Number analyzed (Participants) | 19 | 33 | 2
g/cm^2
  Neck of Femur (Month 24- Week 2) | 0.2 (0.91) | -0.1 (0.06) | -0.1 (0.05)
  Lumbar Spine (Month 24 - Week 2) | -0.0 (0.14) | -0.1 (0.10) | -0.0 (0.07)

ADVERSE EVENTS:
Time Frame: 36 months
Description: Safety set includes all patients in whom transplantation was performed and treated with at least one dose of study drug,had at least one safety assessment after randomization. One patient mis-randomised to "CNI withdrawal" arm but treated in control regimen (CNI+MPA+Steroid), evaluated for safety in control arm.
Arm/Group | Calcineurin Inhibitor (CNI) Withdrawal | CNI+MPA+ Steroid | Steroid Withdrawal
Serious Adverse Events (participants affected / at risk) | 33/48 | 36/48 | 16/30
Other Adverse Events (participants affected / at risk) | 47/48 | 48/48 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Calcineurin Inhibitor (CNI) Withdrawal (N=48) | CNI+MPA+ Steroid (N=48) | Steroid Withdrawal (N=30)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Ileitis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Cyst (General disorders) | 0 | 1 | 0
Device occlusion (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 0 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 4 | 4 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 7 | 4 | 1
Abscess intestinal (Infections and infestations) | 0 | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Bacterascites (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 1 | 0
Cytomegalovirus oesophagitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0
Fungal peritonitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 4 | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Perinephric abscess (Infections and infestations) | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 2 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Salmonellosis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 3 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 2 | 0
Varicella (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0
Wound infection (Infections and infestations) | 2 | 3 | 1
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 0 | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Graft loss (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 2 | 1
Blood creatinine increased (Investigations) | 7 | 4 | 3
Blood pressure increased (Investigations) | 1 | 0 | 0
Drug level above therapeutic (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 1
Urine output decreased (Investigations) | 2 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Glomerular vascular disorder (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 4 | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 3 | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 1 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 2
Haematoma (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 3 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 1 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 1
Lymphocele (Vascular disorders) | 2 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Calcineurin Inhibitor (CNI) Withdrawal (N=48) | CNI+MPA+ Steroid (N=48) | Steroid Withdrawal (N=30)
Anaemia (Blood and lymphatic system disorders) | 15 | 13 | 7
Leukopenia (Blood and lymphatic system disorders) | 2 | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 1
Arrhythmia (Cardiac disorders) | 0 | 2 | 2
Bradycardia (Cardiac disorders) | 2 | 4 | 0
Palpitations (Cardiac disorders) | 4 | 3 | 1
Tachycardia (Cardiac disorders) | 4 | 5 | 1
Cushingoid (Endocrine disorders) | 1 | 3 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 4 | 0
Vision blurred (Eye disorders) | 1 | 4 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 7 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 5 | 0
Constipation (Gastrointestinal disorders) | 22 | 29 | 15
Diarrhoea (Gastrointestinal disorders) | 19 | 12 | 5
Dyspepsia (Gastrointestinal disorders) | 7 | 2 | 0
Epigastric discomfort (Gastrointestinal disorders) | 2 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 8 | 1
Mouth ulceration (Gastrointestinal disorders) | 6 | 3 | 3
Nausea (Gastrointestinal disorders) | 24 | 19 | 7
Paraesthesia oral (Gastrointestinal disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 14 | 16 | 4
Chest discomfort (General disorders) | 1 | 4 | 0
Chest pain (General disorders) | 3 | 8 | 2
Oedema (General disorders) | 8 | 8 | 4
Oedema peripheral (General disorders) | 21 | 17 | 3
Pain (General disorders) | 5 | 6 | 0
Pyrexia (General disorders) | 6 | 8 | 6
Transplant rejection (Immune system disorders) | 7 | 5 | 0
Cellulitis (Infections and infestations) | 3 | 3 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 1
Herpes simplex (Infections and infestations) | 0 | 3 | 0
Herpes zoster (Infections and infestations) | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 1 | 8 | 2
Oral candidiasis (Infections and infestations) | 3 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 9 | 22 | 3
Urinary tract infection (Infections and infestations) | 13 | 15 | 6
Wound infection (Infections and infestations) | 3 | 4 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 13 | 5 | 6
Contusion (Injury, poisoning and procedural complications) | 2 | 4 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 2 | 5 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 4 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 0 | 4 | 1
Procedural pain (Injury, poisoning and procedural complications) | 14 | 11 | 2
Skin laceration (Injury, poisoning and procedural complications) | 2 | 4 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 7 | 1
Wound complication (Injury, poisoning and procedural complications) | 10 | 6 | 4
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 4 | 6 | 1
Alanine aminotransferase increased (Investigations) | 4 | 0 | 0
Blood cholesterol increased (Investigations) | 2 | 4 | 1
Blood creatinine increased (Investigations) | 12 | 13 | 7
Blood glucose increased (Investigations) | 4 | 5 | 2
Blood magnesium decreased (Investigations) | 3 | 0 | 0
Blood phosphorus decreased (Investigations) | 5 | 1 | 2
Hepatic enzyme increased (Investigations) | 3 | 3 | 2
Urine output decreased (Investigations) | 9 | 13 | 7
Weight increased (Investigations) | 8 | 6 | 2
White blood cell count decreased (Investigations) | 1 | 4 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 5 | 4
Fluid overload (Metabolism and nutrition disorders) | 4 | 10 | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 6 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 12 | 9 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 10 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 11 | 15 | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 10 | 9 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 10 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 7 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 7 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 5 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 9 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 9 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 1
Dizziness (Nervous system disorders) | 8 | 10 | 2
Headache (Nervous system disorders) | 10 | 19 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 4 | 0
Lethargy (Nervous system disorders) | 5 | 6 | 0
Paraesthesia (Nervous system disorders) | 6 | 1 | 0
Tremor (Nervous system disorders) | 3 | 8 | 1
Anxiety (Psychiatric disorders) | 3 | 6 | 0
Depression (Psychiatric disorders) | 3 | 2 | 1
Insomnia (Psychiatric disorders) | 10 | 8 | 3
Bladder spasm (Renal and urinary disorders) | 6 | 2 | 4
Dysuria (Renal and urinary disorders) | 5 | 8 | 6
Haematuria (Renal and urinary disorders) | 8 | 7 | 4
Hydronephrosis (Renal and urinary disorders) | 3 | 2 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 3
Polyuria (Renal and urinary disorders) | 2 | 6 | 0
Renal tubular necrosis (Renal and urinary disorders) | 6 | 2 | 4
Menorrhagia (Reproductive system and breast disorders) | 4 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 12 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 4 | 4
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1 | 6 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 6 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Hypertension (Vascular disorders) | 24 | 22 | 10
Hypotension (Vascular disorders) | 7 | 9 | 1
Lymphocele (Vascular disorders) | 3 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.